CLINICAL TRIAL: NCT02604199
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Multi-dose Study to Determine the Depth of Hepatitis B Surface Antigen (HBsAg) Reduction Following Intravenous ARC-520 in Combination With Entecavir or Tenofovir in Patients With HBeAg Negative, Chronic Hepatitis B Virus (HBV) Infection
Brief Title: A Multi-dose Study of ARC-520 in Patients With Hepatitis B 'e' Antigen (HBeAg) Negative, Chronic Hepatitis B Virus (HBV) Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision to discontinue trial
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Heparc-2002; 2014-004145-27 (EudraCT Number)
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — ARC-520; entecavir; Tenofovir; Histamine Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PBO Low Dose (Placebo Comparator): 0.9% normal saline, once every 4 weeks for 4 doses plus daily oral entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg) throughout the study period
  Interventions: Other: placebo; Drug: entecavir; Drug: tenofovir; Drug: antihistamine
- PBO High Dose (Placebo Comparator): 0.9% normal saline, once every 4 weeks for 4 doses plus daily oral entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg) throughout the study period
  Interventions: Other: placebo; Drug: entecavir; Drug: tenofovir; Drug: antihistamine
- ARC-520 Injection 1 mg/kg (Experimental): Intravenous ARC-520 at 1.0 mg/kg, once every 4 weeks for 4 doses plus daily oral entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg) throughout the study period
  Interventions: Drug: ARC-520 Injection; Drug: entecavir; Drug: tenofovir; Drug: antihistamine
- ARC-520 Injection 2 mg/kg (Experimental): Intravenous ARC-520 at 2.0 mg/kg, once every 4 weeks for 4 doses plus daily oral entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg) throughout the study period
  Interventions: Drug: ARC-520 Injection; Drug: entecavir; Drug: tenofovir; Drug: antihistamine

INTERVENTIONS:
Drug: ARC-520 Injection — ARC-520 Injection was administered concomitantly, IV with 0.9% normal saline using an infusion rate of 0.4 mL/min for study treatment and 3.6 mL/min for saline.
  Arms: ARC-520 Injection 1 mg/kg; ARC-520 Injection 2 mg/kg
Other: placebo — Placebo was administered concomitantly, IV with 0.9% normal saline using an infusion rate of 0.4 mL/min for study treatment and 3.6 mL/min for saline.
  Arms: PBO High Dose; PBO Low Dose
Drug: entecavir — All participants will take entecavir or tenofovir throughout the study. Participants will be instructed to take their medication daily.
Drug: tenofovir — All participants will take entecavir or tenofovir throughout the study. Participants will be instructed to take their medication daily.
Drug: antihistamine — All participants will be pretreated with an oral antihistamine, administered 2 hours (±30 minutes) pre-dose. The antihistamine used should in general be an H1>H2 receptor blocker and would include diphenhydramine 50 mg, cetirizine 10 mg, chlorpheniramine 8 mg or hydroxyzine 50 mg. The Investigator is free to choose any of these antihistamines available locally and consistent with their country's Marketing Authorisation.

SUMMARY:
Patients with chronic HBV infection will receive either ARC-520 or placebo in combination with entecavir or tenofovir, and be evaluated for safety and efficacy.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, multi-dose study of ARC-520 in combination with entecavir or tenofovir administered to patients with Hepatitis B 'e' Antigen (HBeAg) negative and immune active chronic HBV infection. Eligible patients who have signed an Ethics Committee - approved informed consent, will be enrolled and will receive ARC-520 or placebo in combination with entecavir or tenofovir. The study will enroll up to a total of 60 eligible chronic HBV infected patients. Patients will undergo the following evaluations at regular intervals during the study: medical history, physical examinations, vital sign measurements (blood pressure, heart rate, respiratory rate and temperature), weight, adverse events assessment (AEs), 12-lead electrocardiograms (ECGs), liver fibrosis testing, concomitant medication assessment, blood sample collection for hematology, coagulation,chemistry, lactate, Pharmacokinetic (PK) measures (in a subset of patients), exploratory Pharmacodynamic (PD) measures, urinalysis, HBV serology, Follicle Stimulating Hormone (FSH) testing (post-menopausal females) and pregnancy testing for females of childbearing potential. Clinically significant changes including AEs will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the patient is lost to follow-up. For each patient, the duration of the study is approximately 33 weeks from screening to the Day 169 follow-up visit. For patients enrolling into a planned extension study, the total duration of this study is approximately 25 weeks from screening to Day 113 end of study visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 75 years of age
* Written informed consent
* No clinically significant abnormalities at screening/pre-dose 12-lead ECG assessment
* No new abnormal finding of clinical relevance at the screening evaluation.
* Diagnosis of HBeAg negative, immune active, chronic HBV infection
* > 2 months of continuous treatment with daily, oral entecavir or tenofovir
* Willingness to continue taking entecavir or tenofovir throughout the study.
* Must use 2 effective methods of contraception (double barrier contraception or hormonal contraceptive along with a barrier contraceptive) (both male and female partners)

Exclusion Criteria:

* Pregnant or lactating
* Acute signs of hepatitis/other infection within 4 weeks of screening
* Antiviral therapy other than entecavir or tenofovir within 3 months of screening
* Prior treatment with interferon in the last 3 years.
* Use within the last 6 months or anticipated requirement for anticoagulants, corticosteroids, immunomodulators, or immunosuppressants.
* Use of prescription medication within 14 days prior to treatment administration except: topical products without systemic absorption, statins (except rosuvastatin), hypertension medications, or hormonal contraceptives.
* Depot injection or implant of any drug within 3 months prior to treatment administration, except injectable/implantable birth control.
* Diagnosis of diabetes mellitus.
* History of autoimmune disease especially autoimmune hepatitis.
* Human immunodeficiency virus (HIV) infection.
* Sero-positive for Hepatitis C Virus (HCV), and/or a history of delta virus hepatitis.
* Hypertension defined as blood pressure > 150/100 mmHg
* History of cardiac rhythm disturbances
* Family history or congenital long QT syndrome, Brugada syndrome or unexplained sudden cardiac death
* Symptomatic heart failure, unstable angina, myocardial infarction, severe cardiovascular disease within 6 months prior to study entry.
* History of malignancy except for adequately treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, or in situ cervical cancer.
* Has had a major surgery within 3 months of screening.
* History of alcohol and/or drug abuse < 12 months from screening.
* Regular uses of alcohol within 6 months prior to screening (ie, more than 14 units of alcohol per week).
* Evidence of severe systemic acute inflammation, sepsis, or hemolysis.
* Diagnosed with a significant psychiatric disorder.
* Use of recreational drugs, such as marijuana, within 3 months prior to screening
* Use of drugs such as cocaine, phencyclidine (PCP), and methamphetamines, within 1 year prior to screening.
* History of allergy to bee sting.
* Use of investigational agents or devices within 30 days prior to planned study dosing or current participation in an investigational study.
* Clinically significant history or presence of any gastrointestinal pathology, unresolved gastrointestinal symptoms, liver or kidney disease.
* Presence of cholangitis, cholecystitis, cholestasis, or duct obstruction.
* Clinically significant history or presence of poorly controlled/uncontrolled systemic disease.
* History of fever within 2 weeks of screening.
* Immunized with a live attenuated vaccine within 7 days prior to dosing or planned vaccination (excluding flu vaccine by injection).
* Presence of any medical or psychiatric condition or social situation that impacts compliance or results in additional safety risk.
* Participated in excessive exercise/physical activity within 7 days of screening or planned during the trial.
* History of coagulopathy/stroke within past 6 months, and/or concurrent anticoagulant medication(s).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- China (2):
  - Research Site 1, Hong Kong
  - Research Site 2, Hong Kong
- Germany (9):
  - Research Site 11, Frankfurt
  - Research Site 9, Hamburg
  - Research Site 8, Hanover
  - Research Site 10, Leipzig
  - Research Site 4, Leipzig
  - Research Site 5, München
  - Research Site 3, Tübingen
  - Research Site 6, Ulm
  - Research Site 7, Würzburg
- South Korea (5):
  - Research Site 13, Busan
  - Research Site 15, Incheon
  - Research Site 14, Seoul
  - Research Site 16, Seoul
  - Research Site 12, Yangsan-si Gyeongnam

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PBO Low Dose | PBO High Dose | ARC-520 Injection 1 mg/kg | ARC-520 Injection 2 mg/kg
Started | 9 | 11 | 17 | 21
Completed | 9 | 8 | 17 | 18
Not Completed | 0 | 3 | 0 | 3
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 2 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PBO Low Dose | PBO High Dose | ARC-520 Injection 1 mg/kg | ARC-520 Injection 2 mg/kg | Total
Number analyzed (Participants) | 9 | 11 | 17 | 21 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (12.10) | 48.7 (9.50) | 45.0 (10.48) | 45.7 (10.48) | 46.2 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 7 | 9 | 19
  Male | 7 | 10 | 10 | 12 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Quantitative Hepatitis B Surface Antigen (Log qHBsAg) at Day 113
Description: Change From Baseline in log qHBsAg at Day 113 in response to multiple doses of ARC-520 versus placebo, using a a mixed effect model for repeated measures (MMRM). Includes parameter baseline as a continuous covariate, and treatment and visit as fixed factors, interaction of treatment and visit, and interaction of parameter baseline and visit.
Time Frame: Baseline, Day 113
Population: Intent to treat population: all participants who received at least 1 dose of study drug and had valid qHBsAg values at baseline and at least one time point on or after the Day 15 visit.
Measure: Least Squares Mean (Standard Error); unit: log IU/mL
Groups:
- Placebo: Placebo (low dose or high dose) 0.9% normal saline, once every 4 weeks for 4 doses plus daily oral entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg) throughout the study period
Arm/Group | Placebo | ARC-520 Injection 1 mg/kg | ARC-520 Injection 2 mg/kg
Number analyzed (Participants) | 15 | 14 | 15
log IU/mL | -0.070 (0.033) | -0.157 (0.036) | -0.379 (0.033)
Statistical Analysis 1: Comparison: Placebo vs ARC-520 Injection 1 mg/kg; Test type: Superiority; p = 0.0810, MMRM — Mixed effect model repeat measurement (MMRM) includes terms of parameter baseline as continuous covariate, and treatment and visit as fixed factors, interaction of treatment and visit, and interaction of parameter baseline and visit; Within-subject covariance is unstructured; LS Mean Difference = -0.086, 95% CI 2-sided [-0.183 to 0.011], Standard Error of Mean 0.048
Statistical Analysis 2: Comparison: Placebo vs ARC-520 Injection 2 mg/kg; Test type: Superiority; p < .0001, MMRM — MMRM includes terms of parameter baseline as continuous covariate, and treatment and visit as fixed factors, interaction of treatment and visit, and interaction of parameter baseline and visit. Within-subject covariance is unstructured; LS Mean Difference = -0.309, 95% CI 2-sided [-0.406 to -0.212], Standard Error of Mean 0.048
Statistical Analysis 3: Comparison: ARC-520 Injection 1 mg/kg vs ARC-520 Injection 2 mg/kg; Test type: Superiority; p < .0001, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.223, 95% CI 2-sided [-0.322 to -0.124], Standard Error of Mean 0.049

2. Secondary Outcome: Change From Baseline in Quantitative Hepatitis B Surface Antigen (Log qHBsAg) Over Time
Description: as for outcome 1
Time Frame: Baseline, Day 15, 29, 43, 57, 71, 85, 99
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: log IU/mL
Arm/Group | Placebo | ARC-520 Injection 1 mg/kg | ARC-520 Injection 2 mg/kg
Number analyzed (Participants) | 18 | 15 | 19
log IU/mL
  Day 15 | 3.297 (0.712) | 3.084 (1.004) | 2.506 (0.844)
  Day 29 | 3.291 (0.694) | 3.098 (0.986) | 2.503 (0.846)
  Day 43: number analyzed (Participants) | 15 | 13 | 17
  Day 43 | 3.188 (0.712) | 3.016 (1.124) | 2.509 (0.836)
  Day 57: number analyzed (Participants) | 17 | 13 | 17
  Day 57 | 3.291 (0.705) | 3.072 (1.061) | 2.329 (0.971)
  Day 71: number analyzed (Participants) | 17 | 14 | 18
  Day 71 | 3.206 (0.663) | 3.051 (1.029) | 2.301 (0.969)
  Day 85: number analyzed (Participants) | 16 | 13 | 15
  Day 85 | 3.309 (0.736) | 2.907 (0.963) | 2.366 (0.862)
  Day 99: number analyzed (Participants) | 16 | 13 | 16
  Day 99 | 3.302 (0.700) | 2.938 (1.055) | 2.360 (0.950)
Statistical Analysis 1: Comparison: Placebo vs ARC-520 Injection 1 mg/kg; Day 15; Test type: Superiority; p = 0.0583, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.089, 95% CI 2-sided [-0.181 to 0.003], Standard Error of Mean 0.046
Statistical Analysis 2: Comparison: Placebo vs ARC-520 Injection 2 mg/kg; Day 15; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.176, 95% CI 2-sided [-0.267 to -0.085], Standard Error of Mean 0.045
Statistical Analysis 3: Comparison: ARC-520 Injection 1 mg/kg vs ARC-520 Injection 2 mg/kg; Day 15; Test type: Superiority; p = 0.0670, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.087, 95% CI 2-sided [-0.181 to 0.006], Standard Error of Mean 0.047
Statistical Analysis 4: Comparison: Placebo vs ARC-520 Injection 1 mg/kg; Day 29; Test type: Superiority; p = 0.0875, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.070, 95% CI 2-sided [-0.151 to 0.011], Standard Error of Mean 0.040
Statistical Analysis 5: Comparison: Placebo vs ARC-520 Injection 2 mg/kg; Day 29; Test type: Superiority; p < .0001, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.179, 95% CI 2-sided [-0.259 to -0.100], Standard Error of Mean 0.040
Statistical Analysis 6: Comparison: ARC-520 Injection 1 mg/kg vs ARC-520 Injection 2 mg/kg; Day 29; Test type: Superiority; p = 0.0099, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.109, 95% CI 2-sided [-0.191 to -0.027], Standard Error of Mean 0.041
Statistical Analysis 7: Comparison: Placebo vs ARC-520 Injection 1 mg/kg; Day 43; Test type: Superiority; p = 0.0017, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.143, 95% CI 2-sided [-0.229 to -0.057], Standard Error of Mean 0.043
Statistical Analysis 8: Comparison: Placebo vs ARC-520 Injection 2 mg/kg; Day 43; Test type: Superiority; p < .0001, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.265, 95% CI 2-sided [-0.349 to -0.180], Standard Error of Mean 0.042
Statistical Analysis 9: Comparison: ARC-520 Injection 1 mg/kg vs ARC-520 Injection 2 mg/kg; Day 43; Test type: Superiority; p = 0.0072, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.122, 95% CI 2-sided [-0.209 to -0.035], Standard Error of Mean 0.043
Statistical Analysis 10: Comparison: Placebo vs ARC-520 Injection 1 mg/kg; Day 57; Test type: Superiority; p = 0.0043, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.118, 95% CI 2-sided [-0.197 to -0.039], Standard Error of Mean 0.039
Statistical Analysis 11: Comparison: Placebo vs ARC-520 Injection 2 mg/kg; Day 57; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.298, 95% CI 2-sided [-0.376 to -0.221], Standard Error of Mean 0.039
Statistical Analysis 12: Comparison: ARC-520 Injection 1 mg/kg vs ARC-520 Injection 2 mg/kg; Day 57; Test type: Superiority; p < .0001, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.181, 95% CI 2-sided [-0.261 to -0.100], Standard Error of Mean 0.040
Statistical Analysis 13: Comparison: Placebo vs ARC-520 Injection 1 mg/kg; Day 71; Test type: Superiority; p = 0.0084, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.132, 95% CI 2-sided [-0.228 to -0.035], Standard Error of Mean 0.048
Statistical Analysis 14: Comparison: Placebo vs ARC-520 Injection 2 mg/kg; Day 71; Test type: Superiority; p < .0001, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.338, 95% CI 2-sided [-0.433 to -0.243], Standard Error of Mean 0.047
Statistical Analysis 15: Comparison: ARC-520 Injection 1 mg/kg vs ARC-520 Injection 2 mg/kg; Day 71; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.206, 95% CI 2-sided [-0.304 to -0.108], Standard Error of Mean 0.049
Statistical Analysis 16: Comparison: Placebo vs ARC-520 Injection 1 mg/kg; Day 85; Test type: Superiority; p = 0.0589, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.096, 95% CI 2-sided [-0.195 to 0.004], Standard Error of Mean 0.050
Statistical Analysis 17: Comparison: Placebo vs ARC-520 Injection 2 mg/kg; Day 85; Test type: Superiority; p < .0001, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.335, 95% CI 2-sided [-0.433 to -0.236], Standard Error of Mean 0.049
Statistical Analysis 18: Comparison: ARC-520 Injection 1 mg/kg vs ARC-520 Injection 2 mg/kg; Day 85; Test type: Superiority; p < .0001, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.239, 95% CI 2-sided [-0.340 to -0.137], Standard Error of Mean 0.050
Statistical Analysis 19: Comparison: Placebo vs ARC-520 Injection 1 mg/kg; Day 99; Test type: Superiority; p = 0.0138, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.132, 95% CI 2-sided [-0.236 to -0.028], Standard Error of Mean 0.052
Statistical Analysis 20: Comparison: Placebo vs ARC-520 Injection 2 mg/kg; Day 99; Test type: Superiority; p < .0001, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.355, 95% CI 2-sided [-0.458 to -0.252], Standard Error of Mean 0.051
Statistical Analysis 21: Comparison: ARC-520 Injection 1 mg/kg vs ARC-520 Injection 2 mg/kg; Day 99; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean = -0.223, 95% CI 2-sided [-0.329 to -0.117], Standard Error of Mean 0.053

3. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), Deaths and Discontinuations Due to AEs
Description: An AE is any untoward medical occurrence which does not necessarily have a causal relationship with this treatment. An SAE is any AE that: results in death; is life-threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is a medically important event or reaction. A treatment emergent AE (TEAE) was defined as an AE that was not present prior to the first study medication administration and started at/after the time of initiation of administration of study medication, or an AE which was present prior to initiation of study medication administration, which increased in severity after study medication administration.
Time Frame: Through Day 169
Population: Safety Population: all participants who received at least 1 dose of study treatment or placebo, and had at least 1 post-dose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | PBO Low Dose | PBO High Dose | ARC-520 Injection 1 mg/kg | ARC-520 Injection 2 mg/kg
Number analyzed (Participants) | 9 | 11 | 17 | 21
Participants
  ≥ 1 AE | 4 | 5 | 6 | 12
  ≥ 1 TEAE | 4 | 4 | 6 | 12
  ≥ 1 Serious TEAE | 0 | 0 | 2 | 1
  Deaths | 0 | 0 | 0 | 0
  ≥ 1 TEAE Leading to Study Discontinuation | 0 | 0 | 0 | 0
  ≥ 1 TEAE Leading to Treatment Discontinuation | 0 | 0 | 0 | 0

4. Secondary Outcome: Pharmacokinetics of ARC-520: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: Due to the early suspension and termination of the study, all pharmacokinetic analyses were removed from the initial statistical analysis plan for this study. No collected samples were analyzed and all were destroyed.
Arm/Group | PBO Low Dose | PBO High Dose | ARC-520 Injection 1 mg/kg | ARC-520 Injection 2 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Pharmacokinetics of ARC-520: Area Under the Plasma Concentration-Time Curve From Time 0 to the Last Quantifiable Plasma Concentration (AUClast)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: as for outcome 4
Arm/Group | PBO Low Dose | PBO High Dose | ARC-520 Injection 1 mg/kg | ARC-520 Injection 2 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Pharmacokinetics of ARC-520: Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUCinf)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: as for outcome 4
Arm/Group | PBO Low Dose | PBO High Dose | ARC-520 Injection 1 mg/kg | ARC-520 Injection 2 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Pharmacokinetics of ARC-520: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: as for outcome 4
Arm/Group | PBO Low Dose | PBO High Dose | ARC-520 Injection 1 mg/kg | ARC-520 Injection 2 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Pharmacokinetics of ARC-520: Clearance (CL)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: as for outcome 4
Arm/Group | PBO Low Dose | PBO High Dose | ARC-520 Injection 1 mg/kg | ARC-520 Injection 2 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Pharmacokinetics of ARC-520: Apparent Volume of Distribution (V)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: as for outcome 4
Arm/Group | PBO Low Dose | PBO High Dose | ARC-520 Injection 1 mg/kg | ARC-520 Injection 2 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Pharmacokinetics of ARC-520: Terminal Elimination Rate Constant (Kel)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: as for outcome 4
Arm/Group | PBO Low Dose | PBO High Dose | ARC-520 Injection 1 mg/kg | ARC-520 Injection 2 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Pharmacokinetics of ARC-520: Terminal Elimination Half-Life (t1/2)
Time Frame: Through 48 hours post-dosing on Day 1 and Day 85
Population: as for outcome 4
Arm/Group | PBO Low Dose | PBO High Dose | ARC-520 Injection 1 mg/kg | ARC-520 Injection 2 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through Day 169
Arm/Group | PBO Low Dose | PBO High Dose | ARC-520 Injection 1 mg/kg | ARC-520 Injection 2 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 2/17 | 1/21
Other Adverse Events (participants affected / at risk) | 4/9 | 4/11 | 4/17 | 8/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PBO Low Dose (N=9) | PBO High Dose (N=11) | ARC-520 Injection 1 mg/kg (N=17) | ARC-520 Injection 2 mg/kg (N=21)
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PBO Low Dose (N=9) | PBO High Dose (N=11) | ARC-520 Injection 1 mg/kg (N=17) | ARC-520 Injection 2 mg/kg (N=21)
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 2
Influenza like illness (General disorders) | 0 | 0 | 1 | 1
Malaise (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The ARC-520 Injection development program was terminated early for regulatory and business reasons secondary to findings occurring in a non-clinical toxicology study. Program termination was not due to safety findings in humans.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No